CLINICAL TRIAL: NCT05038059
Title: Ethanolic Extract of Sapindus Mukorossi as the Final Endodontic Irrigant.
Brief Title: Ethanolic Extract of Sapindus Mukorrossi as Final Endodontic Irrigant.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, ARAIB TAHIR, MDS trainee operative dentistry, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A_tahir
Record Dates: First submitted 2021-08-25; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Irreversible Pulpitis; Apical Periodontitis; Root Canal Infection
MeSH Terms: conditions — Periapical Periodontitis | interventions — Edetic Acid

STUDY DESIGN:
Intervention Model Description: 3 groups assigned 2 with interventions and 1 control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Ethylene diammine tetra acetic acid group (Active Comparator): samples will be rinsed with ethylene diamine tetra acetic acid group, which is the gold standard for final rinse and compares with the experimental group.
  Interventions: Drug: ethylene diamine tetra acetic acid
- 2. Control group (No Intervention): no final irrigant will be used and evaluate the outcomes
- 3. Experimental group (Experimental): final irrigation of root canal will be done with ethanolic extract of sapindus mukorossi
  Interventions: Drug: ethanolic extract of sapindus mukorossi

INTERVENTIONS:
Drug: ethanolic extract of sapindus mukorossi — ethanolic extract will be used as final endodontic irrigant during root canal procedures in extracted teeth.
  Other Names: extract of soapnut
  Arms: 3. Experimental group
Drug: ethylene diamine tetra acetic acid — used as final endodontic irrigant in root canal therapy
  Other Names: edta
  Arms: 1. Ethylene diammine tetra acetic acid group

SUMMARY:
The chief aim of root canal treatment is to reduce the microbial content and prevent further recontamination in the canal. Properly cleaned, shaped and obturated teeth will be having fewer chances of treatment failure. Every tooth has variable, complex canal anatomy consisting of ramifications and lateral canal. The instrumentation alone cannot reach all the areas for cleaning. For proper cleaning and removal of all microorganisms, the canal should be irrigated with any biocompatible, lubricant and antimicrobial agent. An irrigant should have a high compatibility factor, with canals, with obturating material and sealer. It should remove all the superficial barriers from canal tubules and allow sealer penetration, which aids in better adhesion and decreases the chances for recontamination.

Objectives: This study aims to compare the effect of experimental endodontic irrigant Sapindus mukorossi with 17% EDTA, on the microleakage, sealer penetration and interaction with sodium hypochlorite.

Ninety single-rooted teeth will be allocated into 2 experimental groups and a control group of 30 teeth each. The endodontic procedure will be done with protaper files. The sample in group 1 will be irrigated with 3.0% NaOCl after that by 17% EDTA and the sample in group 2 final irrigation will be given with Ethanolic extract of Sapindus mukorossi. After the preparation and final irrigation of all teeth, sterile saline will be used to flush all canals and dried using paper points. Obturation will be done with lateral condensation by gutta-percha. Teeth will be incubated at 37ºc and 100% humidity for 7 days. Varnish will be applied on the root surface except for apical 3mm. The teeth will be sectioned longitudinally and examined at 2 and 5mm from the root apex. The maximum depth of sealer penetration will be measured using a scanning electron microscope and microleakage will be tested through a dye penetration method under a stereomicroscope.

Testing of interaction between irrigant and hypochlorite will be done by placing 1ml irrigant with 1 ml sodium hypochlorite in a round bottom test tube and left for 1 week at 37ºc. An independent observer will look for precipitation formation or color changes

DETAILED DESCRIPTION:
Preparation of ethanolic extract of S.mukorossi:

The desiccated fruit of Sapindus mukorossi will be used for the formulation of an experimental root canal irrigant. The dry pericarps of s. mukorossi (≈ 1.0 kg) which is present around the seed nut, will be separated with a sharp blade. These pericarps will be blended to produce fine particles in a sterilized home blender (Enviro 3 in 1 juicer blender ENJ301). The resultant 10gram powder will be soaked in 100ml of absolute ethanol (99%) for 24hours at normal room temperature. This solvent will be filtered and removed with help of a rotary evaporator, and extract will be kept in cleaned screw-capped vials (Premium Vials B4702-12 Glass with Screw Cap) at -20º C until use. To form an operational concentration of 5 mg/ml, the extract will be re-dissolved in distilled water.

All samples were prepared by a single operator using the following protocol. After extraction tooth was stored in 0.1% thymol. Until further use. Specimens were randomly divided into 3 groups through computer-generated software. There will be 30 teeth in each group.

Chamber opening was done with # 4 diamond cutting round bur, a #10 K-type file (Maillefer/Dentsply) was introduced into each root canal till it could be seen outside the apical foramen. The working length will be decided by decreasing this length by 1mm. A single operator using K-type files (Maillefer/Dentsply) initially than with the ProTaper Universal System (Dentsply-Maillefer) up to F2 was performed. Irrigation was performed at each change of file with 2.5mL of 3% NaOCl (canasol). After instrumentation the sample Group 1 would be irrigated with 3ml of 17% EDTA and left in the canal for 1 minute. Group 2 will be irrigated with Sapindus mukorossi finally all groups will be flushed with 5ml of 0.9% normal saline. The control group's final irrigation was done with 0.9% saline.

Afterward, the specimen was dried with F2 sterile absorbent paper points and an F2 gutta-percha cone was selected as the master cone. Sealapex (Sybron-Endo, Glendora, CA, USA) sealer was mixed according to the manufacturer's instructions and placed in the canal via the help of a 25# k file.

* Mastercone was inserted up to the working length and tug back was assessed.
* Sealer application was performed in the manner described above.
* The GP was inserted up to the working length after the apical 2mm of the master cone was evenly coated with the sealer.
* The finger spreaders #25 and #20 (MANI, Japan) were placed into the canal to make room for the accessory GP.
* The process was repeated until the #20 spreader was unable to enter the canal's coronal one-third.
* Excess GP was seared off using a hot condenser, and coronal GP was vertically compacted to produce a good coronal seal.
* The access cavity was sealed with GIC restorative type(3M, ESPE) All samples were stored in an incubator (binder GmbH, Germany) at 37oc under 100% humidity for 1 week, to allow for the sealer to set completely.

3.10.1 Preparation of the sample for stereomicroscopic analysis of dye penetration: After the samples were retrieved from the incubator they were allowed to air dry for 10 minutes. All samples in the experimental group were coated with two layers of colored nail varnish, except the apical 2mm of the root apex.

After complete drying of nail varnish, the roots were then vertically placed in 1% methylene blue dye (WellcoSol, TM) for 72hours.

After 3 days, the samples were washed for 5 minutes under running tap water and left to air dry fully. To avoid dye introduction onto the inner root surface during sectioning, nail polish and dye were scraped off the samples with a scalpel and surgical blade #15 (Bisturi Ucu, Turkey). The tooth was cut in half longitudinally, parallel to its long axis. To ensure that the sectioning was performed through the center of the root and to prevent damage to the obturated canal space, 2mm deep longitudinal grooves were placed in the center of the buccal and lingual root surface using a diamond disc in a slow-speed handpiece (Nakanishi Inc (NSK), Japan), with caution not to invade the canal space. The teeth were then fractured longitudinally with a double tapered chisel and a mallet, preserving the entire obturation space.

The samples were then viewed under Stereiomicroscope (Olympus VM-ILA-2) in the bioinformatics and Molecular Medicine Laboratory (DRIBBS, DUHS) under 30x magnification. The images were captured and uploaded to IMAGE J software (National Institute of Health, USA). The samples were examined by two blinded observers (endodontists). The investigator determined apical microleakage by measuring the linear depth of dye penetration, which is defined as the maximum dye penetration distance from the root apex to the coronal extent. In the performa, all measures were measured in millimeters (mm).

For dentinal tubule penetrance:

Another half of the tooth was left to desiccate for 24 hours in 40-100% ethyl alcohol. Then specimen will be mounted on metallic stubs and gold-sputtered. Under an electron microscope, a photomicrograph will be taken. Samples were studied for dentinal tubule penetration of sealers at two levels - 2 and 5mm from the root apex by two independent observer's reliability will be checked. Photomicrographs showing the maximum penetration at each level were taken. The distance of the points was measured from the sealer-dentin interface and the depth of penetration was calculated.

For interaction with sodium hypochlorite:

For the assessment of precipitate formation, solutions of 17% EDTA, S.mukorossi, and 3% NaOCl will be used. Each polystyrene round-bottom tube (Falcon; Thermo Fischer Scientific, Waltham, MA) will be filled with 2mL extract of S. mukorossi and17% EDTA respectively. Tube 3 will be filled with a mixture of 1 mL of S.mukorossi and 1 mL 3% NaOCl. Tube 4 was filled with 17% EDTA with NaoCl. Left on 95% humidity at 37ºC for 1 week. An unbiased observer was observing every tube for precipitate formation after every 15minutes for first 2 hours and at 24-hour intervals for 1 week. To avoid any error this procedure repeated 3 times

ELIGIBILITY:
Inclusion Criteria:

* Extracted single rooted teeth with mature apices. (carious/ non carious)
* Teeth extracted for orthodontic and periodontal purpose.
* Patient age between 18 to 40 years.

Exclusion Criteria:

* Intracanal calcification. (will be assessed from pre-operative radiograph before extraction)
* Root dilacerations.
* Root caries, fracture or cracked.
* Root resorption.
* Previously treated or initiated root canal treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
microleakage | in a month
  measured in milimeter by steriomicroscope
dentinal tubule penetration of selaer | 2 months
  measured in micrometer by scanning electron microscope
interaction of extract of sapindus mukorossi with hypochlorite | in 4 weeks
  precipitate formation visible with naked eye

CONTACTS AND LOCATIONS:
Overall Officials: Araib AT Tahir, BDS, Principal Investigator — dow university
Locations (1):
- Dr. Araib Tahir, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Thaha KA, Varma RL, Nair MG, Sam Joseph VG, Krishnan U. Interaction between Octenidine-based Solution and Sodium Hypochlorite: A Mass Spectroscopy, Proton Nuclear Magnetic Resonance, and Scanning Electron Microscopy-based Observational Study. J Endod. 2017 Jan;43(1):135-140. doi: 10.1016/j.joen.2016.09.015. Epub 2016 Dec 6. PMID 27939737
- [Background] Pommel L, About I, Pashley D, Camps J. Apical leakage of four endodontic sealers. J Endod. 2003 Mar;29(3):208-10. doi: 10.1097/00004770-200303000-00011. PMID 12669883
- [Background] Farhad AR, Barekatain B, Koushki AR. The Effect of Three Different Root Canal Irrigant Protocols for Removing Smear Layer on the Apical Microleakage of AH26 Sealer. Iran Endod J. 2008 Summer;3(3):62-7. Epub 2008 Jul 10. PMID 24146672
- [Background] Violich DR, Chandler NP. The smear layer in endodontics - a review. Int Endod J. 2010 Jan;43(1):2-15. doi: 10.1111/j.1365-2591.2009.01627.x. PMID 20002799
- [Background] Bloomfield SF, Miles GA. The antibacterial properties of sodium dichloroisocyanurate and sodium hypochlorite formulations. J Appl Bacteriol. 1979 Feb;46(1):65-73. doi: 10.1111/j.1365-2672.1979.tb02582.x. No abstract available. PMID 35510
- [Background] Kuci A, Alacam T, Yavas O, Ergul-Ulger Z, Kayaoglu G. Sealer penetration into dentinal tubules in the presence or absence of smear layer: a confocal laser scanning microscopic study. J Endod. 2014 Oct;40(10):1627-31. doi: 10.1016/j.joen.2014.03.019. Epub 2014 May 10. PMID 25260735